CLINICAL TRIAL: NCT01416428
Title: Phase 1b/2, Multicenter, Open-label Study of the Safety and Activity of Oprozomib in Patients With Hematologic Malignancies
Brief Title: Open-label Study of the Safety and Activity of Oprozomib in Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A program evaluation identified that the safety profile and pharmacokinetic (PK) characteristics of the formulation used in all oprozomib studies required further optimization and thus enrollment in 2011-001 was halted.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-001
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma; Waldenstrom Macroglobulinemia
Keywords: multiple myeloma; waldenstrom macroglobulinemia
MeSH Terms: conditions — Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — ONX 0912

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QDx2 Dosing Schedule (Experimental): QDx2 is defined as patients receiving Oprozomib Tablets once daily on Days 1, 2, 8, and 9 of the 14-day cycle.
  The schedule will be evaluated in Phase 1 for MTD in patients with hematologic malignancies, and will also be evaluated in Phase 2 for ORR in patients with MM and WM.
  Interventions: Drug: oprozomib
- QDx5 Dosing Schedule (Experimental): QDx5 is defined as patients receiving Oprozomib Tablets once daily on Days 1 to 5 of the 14-day cycle.
  The schedule will be evaluated in Phase 1 for MTD in patients with hematologic malignancies, and will also be evaluated in Phase 2 for ORR in patients with MM and WM.
  Interventions: Drug: oprozomib

INTERVENTIONS:
Drug: oprozomib — Patients enrolled will receive Oprozomib Tablets once daily either on Days 1-5 (QDx5 schedule) or on Days 1, 2, 8, and 9 (QDx2 weekly schedule) of the 14-day treatment cycle.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD), activity, and safety of oprozomib in patients with hematologic malignancies.

ELIGIBILITY:
INCLUSION CRITERIA:

Phase 1b

* Histologically confirmed diagnosis of a hematologic malignancy, excluding patients with acute leukemia or MDS.
* Relapsed after standard therapy for their malignancy and considered to be an appropriate candidate for a Phase 1 clinical study by their treating physician.

Phase 2

* Multiple myeloma with measurable disease
* Waldenström macroglobulinemia with symptomatic relapse
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.

Ethical/Other

* Patients must sign a written informed consent form in accordance with federal, local, and institutional guidelines.
* Female patients of childbearing potential must have a negative serum or urine pregnancy test and agree to use effective contraception. Male patients must use an effective barrier method of contraception.

EXCLUSION CRITERIA:

* Chemotherapy with approved or investigational anticancer therapeutics, including steroid therapy intended to treat underlying malignancy, within 3 weeks prior to first dose or 6 weeks for antibody therapy.
* Radiation therapy within 3 weeks prior to first dose. Radioimmunotherapy within 8 weeks prior to first dose. Localized radiation therapy within 1 week prior to first dose.
* Immunotherapy within 3 weeks prior to first dose (except for antibody therapy, where 6 weeks is required).
* Prior stem cell transplant (SCT) therapy (autologous SCT within the prior 8 weeks; allogeneic SCT within the prior 16 weeks). Patients with prior allogeneic SCT should not have evidence of moderate-to-severe graft-vs-host disease (GvHD; as defined in Filipovich 2005).
* Evidence of central nervous system (CNS) lymphoma.
* Prior treatment with carfilzomib unless in the phase 2.
* Major surgery within 3 weeks prior to first dose.
* Symptomatic Congestive heart failure, ischemia, conduction abnormalities, or myocardial infarction within 6 months.
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals.
* Known or suspected human immunodeficiency virus (HIV) infection or patients who are HIV seropositive.
* Active hepatitis A, B, or C infection.
* Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose.
* Patients with pleural effusions requiring routine thoracentesis or ascites requiring routine paracentesis.
* History of previous clinically significant GI bleed in the last 6 months prior to first dose.
* Female patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-10-15 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Determine the MTD (Phase 1) and ORR (Phase 2). | 6 weeks to 18 months
  Phase 1- Determine Maximum Tolerated Dose (MTD) with 3 + 3 Dose Escalation Cohorts in patients hematologic malignancies.
  Phase 2- The Phase 2 portion of this trial will enroll patients with Multiple Myeloma (MM) and Waldenstrom Macroglobulinemia (WM) into separate arms to assess activity of oprozomib in these patient groups. The purpose of the Phase 2 portion of the study is to estimate the best ORR (for each group separately).

SECONDARY OUTCOMES:
Evaluate the duration of response (DOR) | 64 months
  Duration of Response is defined as the time from first evidence of partial response (PR) or better to confirmation of disease progression or death due to any cause.
Estimate the clinical benefit response (CBR) | 64 months
  CBR is defined as Overall Response Rate (ORR) plus Minimal Response (MR) of oprozomib in patients with multiple myeloma (MM)
Estimate the major response for Waldenström macroglobulinemia (WM) | 64 months
  Major response for WM subjects is defined as Complete Response (CR) plus Very Good Partial Response (VGPR) plus Partial Response (PR). Major response to be equal or greater than (PR)
Evaluate progression-free survival (PFS) for multiple myeloma (MM) subjects | 64 months
  Progression-Free Survival is defined as the time from the start of treatment to disease progression or death (due to any cause), whichever comes first
Evaluate the PFS for Waldenström macroglobulinemia (WM) subjects | 64 months
  Progression-Free Survival is defined as the time from the start of treatment to disease progression or death (due to any cause), whichever comes first
PK parameters - maximum plasma concentration (Cmax) | 55 months
  PK analyses to be performed on oprozomib and its metabolite(s) concentrations in order to estimate the maximum observed drug concentration (Cmax) value after oral administration
PK parameters - time of maximum plasma concentration (tmax) | 55 months
  PK analyses to be performed on oprozomib and its metabolite(s) concentrations in order to estimate the time to reach Cmax (tmax)
PK parameters - plasma concentration-time curve (AUC) | 55 months
  PK analyses to be performed on oprozomib and its metabolite(s) concentrations in order to estimate the area under the plasma concentration-time curve
Assess renal elimination of oprozomib and its metabolites (Phase 1b only) | 55 months
  Urine will be collected over 24 hours to assess renal elimination of oprozomib and its metabolites following dosing on Day 1 of Cycle 1 for all patients.
Change from Baseline in hematology laboratory results | 64 months
  Assess the change from baseline in hematology panel
Change from Baseline in serum chemistry results | 64 months
  Assess the change from baseline in serum chemistry panel
Change from Baseline in vital signs | 64 months
  Assess the change from baseline in vital signs including blood pressure, pulse, and temperature
Change from Baseline in weight | 64 months
  Assess the change from baseline in weight
Evaluate safety of oprozomib in Phase 2 | Until 30 days after the end of study (64 months)
  Safety to be defined by incidence, nature, severity, and relatedness of adverse events (AEs), including all serious adverse events (SAEs)
Assess the effect on transfusion/ red blood cell (RBC) growth factor requirements (Phase 2 only) for WM only | 64 months
  Change from Baseline (prior 1 month) transfusion/RBC growth factor requirement in frequency and volume in WM (Phase 2 only)
Assess the effect on plasmapheresis requirements (Phase 2 only) for WM only | 64 months
  Change from Baseline (prior 1 month) plasmapheresis requirement in frequency and volume in WM (Phase 2 only)
Assess the effect on lymphoplasmacytic cells in the bone marrow (Phase 2 only) for WM only | 64 months
  Change from Baseline in percent of lymphoplasmacytic cells in the bone marrow in WM (Phase 2 only)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- United States (19):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Pacific Cancer Care, Salinas, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mass General Hospital, Boston, Massachusetts
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine Division of Oncology, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University, Hackensack, New Jersey
  - Hematology Oncology of Northern New Jersey, Morristown, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Sarah Cannon Research Institute / Tennessee Oncology, PLLC, Nashville, Tennessee
  - Columbia Basin Hematology and Oncology, Kennewick, Washington

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com